CLINICAL TRIAL: NCT01106638
Title: A Trial to Test the Efficacy of a Tailored Intensive Smoking Cessation Intervention in Persons With HIV (PWHs)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: Albert Einstein College of Medicine (Other); Yale University (Other)
Responsible Party: Principal Investigator, Jonathan Shuter, principal investigator, Montefiore Medical Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R21DA023362 (NIH)
Record Dates: First submitted 2010-04-19; First posted 2010-04-20 (Estimated); Last update posted 2018-04-27 (Actual); Status verified 2018-04

CONDITIONS: Smoking; HIV Infections; AIDS
Keywords: HIV; AIDS; Smoking; Tobacco; Cessation; Tobacco use in persons living with HIV/AIDS
MeSH Terms: conditions — Smoking; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intensive behavioral intervention (Experimental): Eight session, behavioral intervention targeting HIV-infected smokers
  Interventions: Behavioral: Positively Smoke Free
- Standard care (Active Comparator): Advice to quit, smoking cessation brochure, offer of nicotine patch
  Interventions: Behavioral: Standard care

INTERVENTIONS:
Behavioral: Positively Smoke Free — An eight session, group therapy intervention targeting smokers living with HIV/AIDS
  Arms: Intensive behavioral intervention
Behavioral: Standard care — Advice to quit, smoking cessation brochure, and offer of nicotine patches
  Arms: Standard care

SUMMARY:
The purpose of this study is to determine whether an intensive, eight session behavioral intervention is superior to standard care in achieving abstinence from cigarettes in smokers living with HIV/AIDS.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infection
* current cigarette smoker
* high motivation to quit

Exclusion Criteria:

* Pregnancy
* breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2009-12 (Actual); Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Three month point-prevalence abstinence from cigarettes | 3 months post-intervention

SECONDARY OUTCOMES:
Three month continuous abstinence from cigarettes | Three months post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Shuter, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

REFERENCES:
- [Derived] Shuter J, Pearlman BK, Stanton CA, Moadel AB, Kim RS, Weinberger AH. Gender Differences among Smokers Living with HIV. J Int Assoc Provid AIDS Care. 2016 Sep;15(5):412-7. doi: 10.1177/2325957416649439. Epub 2016 May 23. PMID 27215559
- [Derived] Moadel AB, Bernstein SL, Mermelstein RJ, Arnsten JH, Dolce EH, Shuter J. A randomized controlled trial of a tailored group smoking cessation intervention for HIV-infected smokers. J Acquir Immune Defic Syndr. 2012 Oct 1;61(2):208-15. doi: 10.1097/QAI.0b013e3182645679. PMID 22732470